CLINICAL TRIAL: NCT00597129
Title: A Phase I, Dose-Escalating Study to Investigate the Safety, Tolerability, Pharmacokinetics and Dosimetry of a Single Dose of 90YHumanized PAM4 IgG in Patients With Locally Advanced/Metastatic Pancreatic Cancer
Brief Title: Safety and Efficacy Study of 90Y-hPAM4 at Different Doses
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: William Wegener, MD, PHD, Immunomedics, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM-T-hPAM4-01; NCT00303680 (obsolete NCT alias)
Record Dates: First submitted 2008-01-08; First posted 2008-01-17 (Estimated); Last update posted 2021-08-19 (Actual); Status verified 2008-01

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer; cancer of the pancreas; pancreas cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — MUC-1 monoclonal antibody

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Multi Dose levels (Experimental): different doses of 90YhPAM4 will be given only once.
  Interventions: Biological: 90Y-hPAM4

INTERVENTIONS:
Biological: 90Y-hPAM4 — Single dose of 90Y-hPAM4 will be given and all patients will be followed for 12 weeks.
  Other Names: 111-IN-hPAM4; MUC-1 antibody

SUMMARY:
Safety study to determine highest dose of 90Y-hPAM4 can be safety administered

DETAILED DESCRIPTION:
radiolabeled anti-MUC1 humanized antibody) administered intravenously as a single dose to patients with locally advanced and/or metastatic pancreatic cancer. The primary objective is to determine the dose-limiting toxicity (DLT) and maximum tolerated dose (MTD) of 90Y-hPAM4 in this population. Secondary objectives include the assessment of tumor targeting, biodistribution, organ dosimetry and pharmacokinetics (PK) of 90Y-hPAM4 as determined by pre-therapy administration of 111In-hPAM4, the assessment of the antigenicity of 90Y-hPAM4, as determined by development of human anti-humanized antibodies (HAHA), and to obtain preliminary information on the efficacy of single dose 90Y-hPAM4 in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, >18 years of age, who are able to understand and give written informed consent.
* Histologically or cytologically confirmed, Stage III or IV pancreatic adenocarcinoma.
* Patients with Stage III (locally advanced) disease must have documented progression after failing primary therapy
* Patients with Stage IV (metastatic) disease must not have received more than one chemotherapy regimen.
* Measurable disease by CT, with at least on lesion >1.5 cm in one dimension.
* Karnofsky performance status > 70 % (Appendix A).
* Expected survival > three months.
* At least 4 weeks beyond chemotherapy, radiotherapy, major surgery, other experimental treatments, and recovered from all acute toxicities.
* At least 2 weeks beyond corticosteroids, except low doses (i.e., 20 mg/day of prednisone or equivalent) to treat nausea or other illness such as rheumatoid arthritis
* Adequate hematology without ongoing transfusional support (hemoglobin > 10 g/dL, ANC > 1,500 per mm3, platelets > 150,000 per mm3)
* Adequate renal and hepatic function (creatinine and bilirubin ≤ 1.5 X IULN, AST and ALT ≤ 2.0 X IULN)
* Otherwise, all toxicity at study entry <Grade 1 by NCI CTC v3.0.

Exclusion Criteria:

* Women who are pregnant or lactating.
* Women of childbearing potential and fertile men unwilling to use effective contraception during study until conclusion of 12-week post-treatment evaluation period.
* Known metastatic disease to the central nervous system.
* Presence of bulky disease (defined as any single mass >10 cm in its greatest dimension)
* Patients with >Grade 2 anorexia, nausea or vomiting, and/or signs of intestinal obstruction.
* Prior treatment with nitrosureas, actinomycin-D, radioimmunotherapy or other antibody-based therapies (murine, chimeric, humanized or human) Prior radiation dose >3,000 cGy to the liver, >2,000 cGy to lungs and kidneys or prior external beam irradiation to a field that includes more than 30% of the red marrow.
* Patients with non-melanoma skin cancer or carcinoma in situ of the cervix are not excluded, but patients with other prior malignancies must have had at least a 5- year disease free interval.
* Patients known to be HIV positive, hepatitis B positive, or hepatitis C positive.
* Known history of active coronary artery disease, unstable angina, myocardial infarction, or congestive heart failure present within 6 months or cardiac arrhythmia requiring anti-arrhythmia therapy.
* Known history of active COPD, or other moderate-to-severe respiratory illness present within 6 months.
* Known autoimmune disease or presence of autoimmune phenomena (except rheumatoid arthritis requiring only low dose maintenance corticosteroids).
* Infection requiring intravenous antibiotic use within 1 week.
* Other concurrent medical or psychiatric conditions that, in the Investigator's opinion, may be likely to confound study interpretation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2004-08; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
safety MTD | over the first 12 weeks, then over 2 years

SECONDARY OUTCOMES:
targeting, biodistribution, organ dosimetry | first 2 weeks
pharmacokinetics (PK), antigenicity, | first 12 weeks
efficacy | over first 12 weeks, then over 2 years

CONTACTS AND LOCATIONS:
Overall Officials: William Wegener, MD, PhD, Study Chair — Gilead Sciences
Locations (4):
- United States (4):
  - Goshen Cancer Center, Goshen, Indiana
  - Nebraska Medical Center, Omaha, Nebraska
  - University of Medicine and Dentistry, Newark, New Jersey
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Gold DV, Karanjawala Z, Modrak DE, Goldenberg DM, Hruban RH. PAM4-reactive MUC1 is a biomarker for early pancreatic adenocarcinoma. Clin Cancer Res. 2007 Dec 15;13(24):7380-7. doi: 10.1158/1078-0432.CCR-07-1488. PMID 18094420
- [Background] Modrak DE, Gold DV, Goldenberg DM. Sphingolipid targets in cancer therapy. Mol Cancer Ther. 2006 Feb;5(2):200-8. doi: 10.1158/1535-7163.MCT-05-0420. PMID 16505092
- [Background] Gold DV, Modrak DE, Ying Z, Cardillo TM, Sharkey RM, Goldenberg DM. New MUC1 serum immunoassay differentiates pancreatic cancer from pancreatitis. J Clin Oncol. 2006 Jan 10;24(2):252-8. doi: 10.1200/JCO.2005.02.8282. Epub 2005 Dec 12. PMID 16344318
- [Background] Modrak DE, Karacay H, Cardillo TM, Newsome G, Goldenberg DM, Gold DV. Identification of a Mu-9 (anti-colon-specific antigen-p)-reactive peptide having homology to CA125 (MUC16). Int J Oncol. 2005 Jun;26(6):1591-6. PMID 15870874
- [Background] Modrak DE, Cardillo TM, Newsome GA, Goldenberg DM, Gold DV. Synergistic interaction between sphingomyelin and gemcitabine potentiates ceramide-mediated apoptosis in pancreatic cancer. Cancer Res. 2004 Nov 15;64(22):8405-10. doi: 10.1158/0008-5472.CAN-04-2988. PMID 15548711
- [Background] Gold DV, Modrak DE, Schutsky K, Cardillo TM. Combined 90Yttrium-DOTA-labeled PAM4 antibody radioimmunotherapy and gemcitabine radiosensitization for the treatment of a human pancreatic cancer xenograft. Int J Cancer. 2004 Apr 20;109(4):618-26. doi: 10.1002/ijc.20004. PMID 14991585
- [Background] Gold DV, Schutsky K, Modrak D, Cardillo TM. Low-dose radioimmunotherapy ((90)Y-PAM4) combined with gemcitabine for the treatment of experimental pancreatic cancer. Clin Cancer Res. 2003 Sep 1;9(10 Pt 2):3929S-37S. PMID 14506191
- [Background] Modrak DE, Gold DV, Goldenberg DM, Blumenthal RD. Colonic tumor CEA, CSAp and MUC-1 expression following radioimmunotherapy or chemotherapy. Tumour Biol. 2003 Jan-Feb;24(1):32-9. doi: 10.1159/000070658. PMID 12743424
- [Background] Reddy PK, Gold DV, Cardillo TM, Goldenberg DM, Li H, Burton JD. Interferon-gamma upregulates MUC1 expression in haematopoietic and epithelial cancer cell lines, an effect associated with MUC1 mRNA induction. Eur J Cancer. 2003 Feb;39(3):397-404. doi: 10.1016/s0959-8049(02)00700-1. PMID 12565994
- [Background] Cardillo TM, Blumenthal R, Ying Z, Gold DV. Combined gemcitabine and radioimmunotherapy for the treatment of pancreatic cancer. Int J Cancer. 2002 Jan 20;97(3):386-92. doi: 10.1002/ijc.1613. PMID 11774294
- [Background] Cardillo TM, Ying Z, Gold DV. Therapeutic advantage of (90)yttrium- versus (131)iodine-labeled PAM4 antibody in experimental pancreatic cancer. Clin Cancer Res. 2001 Oct;7(10):3186-92. PMID 11595713
- [Background] Gold DV, Cardillo T, Goldenberg DM, Sharkey RM. Localization of pancreatic cancer with radiolabeled monoclonal antibody PAM4. Crit Rev Oncol Hematol. 2001 Jul-Aug;39(1-2):147-54. doi: 10.1016/s1040-8428(01)00114-7. PMID 11418312
- [Background] Gold DV, Cardillo T, Vardi Y, Blumenthal R. Radioimmunotherapy of experimental pancreatic cancer with 131I-labeled monoclonal antibody PAM4. Int J Cancer. 1997 May 16;71(4):660-7. doi: 10.1002/(sici)1097-0215(19970516)71:43.0.co;2-e. PMID 9178823
- [Background] Mariani G, Molea N, Bacciardi D, Boggi U, Fornaciari G, Campani D, Salvadori PA, Giulianotti PC, Mosca F, Gold DV, et al. Initial tumor targeting, biodistribution, and pharmacokinetic evaluation of the monoclonal antibody PAM4 in patients with pancreatic cancer. Cancer Res. 1995 Dec 1;55(23 Suppl):5911s-5915s. PMID 7493369
- [Background] Alisauskus R, Wong GY, Gold DV. Initial studies of monoclonal antibody PAM4 targeting to xenografted orthotopic pancreatic cancer. Cancer Res. 1995 Dec 1;55(23 Suppl):5743s-5748s. PMID 7493339
- [Background] Gold DV, Alisauskas R, Sharkey RM. Targeting of xenografted pancreatic cancer with a new monoclonal antibody, PAM4. Cancer Res. 1995 Mar 1;55(5):1105-10. PMID 7866995
- [Background] Gold DV, Lew K, Maliniak R, Hernandez M, Cardillo T. Characterization of monoclonal antibody PAM4 reactive with a pancreatic cancer mucin. Int J Cancer. 1994 Apr 15;57(2):204-10. doi: 10.1002/ijc.2910570213. PMID 7512537